CLINICAL TRIAL: NCT04517435
Title: An Open-Label, Phase I/II Study of ME-401 and R-CHOP in Newly Diagnosed Diffuse Large B-Cell Lymphoma
Brief Title: ME-401 and R-CHOP in Newly Diagnosed Diffuse Large B-Cell Lymphoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Funding unavailable
Sponsor: Deepa Jagadeesh (Other)
Collaborators: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor-Investigator, Deepa Jagadeesh, Principal Investigator, Case Comprehensive Cancer Center
Organization: Case Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE1420
Record Dates: First submitted 2020-08-14; First posted 2020-08-18 (Actual); Results first posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-01

CONDITIONS: Diffuse Large B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — ME-401; Rituximab; Cyclophosphamide; Doxorubicin; Vincristine; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ME-401 + R-CHOP (Experimental): Participants will receive ME-401 dose dependent on dose-escalation schedule at time of enrollment - all will receive standard dose R-CHOP. ME-401 (60 mg) will be given on days 1-4 (dose level 1) OR days 1-7 (dose level 2) of a 21 day cycle with standard dose R-CHOP x 6 cycles.
  Interventions: Drug: ME-401; Drug: Rituximab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisone

INTERVENTIONS:
Drug: ME-401 — ME-401 (60 mg) will be given by mouth every 21 days for 6 cycles on days 1-4 (dose level 1) OR days 1-7 (dose level 2) of a 21 day cycle. Dose escalation will be performed in a standard 3+3 design
  Other Names: PWT-143
Drug: Rituximab — 375 mg/m2 IV/subcutaneous rituximab day 1 of 21-day cycle.
  First dose of rituximab will be given IV and subsequent doses can be either IV or SQ based on institutional guidelines.
  Other Names: Rituxan; Mabthera
Drug: Cyclophosphamide — 750 mg/m2 IV Cyclophosphamide day 1 of 21-day cycle
  Other Names: Cytoxan
Drug: Doxorubicin — 50 mg/m2 IV Doxorubicin day 1 of 21-day cycle
  Other Names: Doxorubicin Hydrochloride
Drug: Vincristine — 1.4 mg/m2 (max 2 mg) IV Vincristine
  Other Names: OncovinTM
Drug: Prednisone — 100mg PO Prednisone Days 1-5 of 21-day cycle

SUMMARY:
This study is being done to evaluate if ME-401 can improve the treatment of patients with diffuse large b-celllymphoma (DLBCL). Many patients with DLBCL that are treated with the standard of care (R-CHOP) are cured. However, a little less than half of patients will have their cancer come back despite being treated. Once DLBCL comes back, it is much harder to treat and treatment is much more aggressive. This study will combine ME-401 with R-CHOP. There are 2 parts to this study: part1 referred to as phase I and part 2 referred to as phase 2. The goal of the phase I study is to find the safest dose to give patients in combination with R-CHOP. The goal of the phase 2 study is to use the safest dose (found in phase 1) in combination with R-CHOP to see if it decreases the rate of cancer coming back after it is treated.

DETAILED DESCRIPTION:
This study is a multi-institution, open-label, phase I/II study designed to evaluate the safety and efficacy of R-CHOP + ME-401 for participants with newly diagnosed DLBCL.

Objectives for the phase I portion of this study are as follows:

Primary objectives:

* To determine the recommended phase 2 dose (RP2D) of ME-401in combination with R-CHOP for participants with newly diagnosed DLBCL.
* To describe tolerability of ME-401 in combination with R-CHOP for participants with newly diagnosed DLBCL.

Objectives for the phase II portion of this study are as follows:

* To estimate the clinical activity of ME-401 in combination with R-CHOP in participants with newly diagnosed DLBCL, as measured by 1 year PFS rate
* To estimate the response rates (complete and partial remission),duration of response (DOR), time to progression (TTP), and overall survival (OS) with ME-401 plus R-CHOP.
* To characterize treatment-related AEs in participants treated with ME-401 plus R-CHOP.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically confirmed diffuse large B-cell lymphoma (DLBCL). Participants with previously diagnosed indolent lymphoma (follicular and marginal zone lymphoma but not small lymphocytic lymphoma) who have transformed to DLBCL are eligible only if they have not previously been treated for indolent lymphoma.

  --If participants received single rituximab (maximum 4-8 doses with no maintenance) for their low grade lymphoma ≥12 months prior to starting study drug are eligible to participate
* Participants must have radiographically measurable disease. At least one bi-dimensionally measurable nodal lesion ≥1.5 cm in its longest diameter by CT scan or MRI, as defined by the Lugano Classification
* Patients participating in the phase II part are allowed to receive brief (<15 days) treatment with glucocorticoids (max dose of prednisone 40 mg) and/or 1 cycle of chemotherapy such as R-CHOP [or some component(s) thereof] for the diagnosis of B-cell lymphoma provided they had all necessary staging tests performed prior to R-CHOPor steroids including CT and/or PET/CTscans, and bone marrow biopsy. Treatment must occur within 30 days prior to enrollment.
* No prior therapy with PI3K inhibitors or Bruton tyrosine kinase (BTK) inhibitors
* ECOG Performance status ≤2. Performance Status of 3 will be accepted if impairment is caused by DLBCL complications and improvement is expected once therapy is initiated.
* Participants must have adequate hematologic, hepatic, and renal function as defined below:

  * Hemoglobin ≥9.0g/dl unless the anemia is clearly due to DLBCL. If there is BM involvement, this criteria can be waived after discussion with the Sponsor Investigator (per investigators discretion).
  * Absolute neutrophil count≥1,000/mcL, unless the neutropenia is clearly due to DLBCL. If there is BM involvement, this criteria can be waived after discussion with the Sponsor Investigator(per investigator discretion)
  * Platelet count ≥75,000/mcl unless thrombocytopenia is clearly due to DLBCL. If there is BM involvement, this criteria can be waived after discussion with the Sponsor Investigator(per investigator discretion)
  * Bilirubin ≤ 2.0 x ULN unless considered secondary to Gilbert's syndrome, in which case ≤ 3 x ULN
  * AST (SGOT) < 2.0 x institutional upper limit of normal
  * ALT (SGPT) < 2.0 x institutional upper limit of normal
  * Creatinine clearance ≥45 mL/min calculated by Cockcroft-Gault or 24 hour collection
* Adequate cardiac function left ventricular ejection fraction (LVEF) ≥50% as assessed by echocardiogram or MUGA (Multi Gated Acquisition Scan).
* QT-interval corrected according to Fridericia's formula (QTcF) ≤450 milliseconds (ms); participants with QTc < 480 msec may be enrolled provided the QTc prolongation is due to a right bundle branch block and stable .
* Negative pregnancy test in women of child-bearing age. The effects of ME-401 on the developing human fetus are unknown. For this reason and because chemotherapeutic agents used in this study are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (double barrier method of birth control or abstinence) 2 weeks prior to initiation of treatment, for the duration of study participation and for 3 months after completing treatment. Should a woman become pregnant or suspect that she is pregnant while she or her partner is participating in this study, she should inform the treating physician immediately. Men must agree to refrain from sperm donation for at least 90 days after the last dose of ME-401
* Participants must have the ability to understand and the willingness to sign a written informed consent document.
* International Prognostic Index must be documented:

  * ECOG performance status ≥2
  * Age ≥60 years
  * extranodal sites ≥ 2
  * LDH >upper limit of normal
  * Ann Arbor Stage III or IV
  * Is there evidence of transformation from indolent lymphoma?

Exclusion Criteria:

* Participants receiving any other investigational agents.
* Known CNS involvement by lymphoma. Participants at high risk for secondary CNS involvement but without neurologic symptoms suspected to be due to lymphoma are allowed to be enrolled and receive prophylactic intrathecal chemotherapy including but not limited to methotrexate, cytarabine and glucocorticoids. Participants who are enrolled and subsequently identified to have pathologic confirmation of CNS involvement by lymphoma may be continued on study at the discretion of the principal investigator.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to R-CHOP.
* Participants with ongoing uncontrolled illness including, but not limited to ongoing significantly active infections requiring intravenous antibiotics, hypertension, angina, arrhythmias, pulmonary disease, or autoimmune dysfunction.
* Uncontrolled autoimmune hemolytic anemia or immune thrombocytopenia.
* Ongoing drug-induced pneumonitis.
* History of clinically significant gastrointestinal (GI) conditions, particularly:

  * Known GI condition that would interfere with swallowing or the oral absorption or tolerance of study drug
  * Pre-existing malabsorption syndrome or other clinical situation that would
* Active congestive heart failure (New York Heart Association [NYHA] Class>2), symptomatic ischemia, or conduction abnormalities uncontrolled by conventional intervention or myocardial infarction within six months prior to enrollment.
* Participants who have tested positive for hepatitis B surface antigen and/or hepatitis B core antibody PLUS have detectable viral load on hepatitis B polymerase chain reaction (PCR) assay (participants with a negative PCR assay are permitted with appropriate anti-viral prophylaxis)
* Positive hepatitis C virus antibody (HCV Ab) participants with positive hepatitis C antibody are eligible if they are negative for hepatitis C virus by PCR
* HIV-positive participants on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with ME-401
* Pregnant or breastfeeding women are excluded from this study because there are no studies assessing the reproductive and developmental toxicity or excretion into breast milk of ME-401. Because there is an unknown, but potential risk for adverse events in nursing infants secondary to treatment of the mother with ME-401, breastfeeding should be discontinued if the mother is treated with ME-401. These potential risks may also apply to other drugs used in this study.
* Other malignancies within the past 3 years except for adequately treated carcinoma of the cervix or basal or squamous cell carcinomas of the skin, or low-risk prostate cancer after curative therapy.
* Participants who have had major surgical procedures or significant traumatic injury within 28 days prior to study treatment.
* Psychiatric illness/social situations that would interfere with study compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-04-28 (Actual); Primary Completion 2023-05-17 (Actual); Study Completion 2023-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deepa Jagadeesh, MD, MPH, Principal Investigator — Cleveland Clinic Taussig Cancer institute, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Taussig Cancer institute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
There are no plans to share individual participant data in order to protect the confidentiality of the subjects who enroll on the study

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I: ME-401 + R-CHOP Dose Level 1: Participants will receive ME-401 dose dependent on dose-escalation schedule at time of enrollment - all will receive standard dose R-CHOP. ME-401 (60 mg) will be given on days 1-4 (dose level 1) of a 21 day cycle with standard dose R-CHOP x 6 cycles.
- Phase I: ME-401 + R-CHOP Dose Level 2; Phase II: ME-401 + R-CHOP: Participants will receive ME-401 dose dependent on dose-escalation schedule at time of enrollment - all will receive standard dose R-CHOP. ME-401 (60 mg) will be given on days 1-7 (dose level 2) of a 21 day cycle with standard dose R-CHOP x 6 cycles.
Period: Overall Study
Arm/Group | Phase I: ME-401 + R-CHOP Dose Level 1 | Phase I: ME-401 + R-CHOP Dose Level 2 | Phase II: ME-401 + R-CHOP
Started | 3 | 6 | 4
Completed | 0 | 0 | 0
Not Completed | 3 | 6 | 4
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Pharmaceutical company discontinued the trial | 3 | 6 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I: ME-401 + R-CHOP Dose Level 1 | Phase I: ME-401 + R-CHOP Dose Level 2 | Phase II: ME-401 + R-CHOP | Total
Number analyzed (Participants) | 3 | 6 | 4 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 1 | 4
  >=65 years | 2 | 4 | 3 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 3 | 7
  Male | 1 | 4 | 1 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 2 | 6 | 4 | 12
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 3 | 6 | 4 | 13
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 6 | 4 | 13

OUTCOME MEASURES:

1. Primary Outcome: Phase I: Number of Clinically Significant Non-hematologic Grade 3 or 4 Treatment-related AEs or Hematologic Grade 3 or 4 Treatment Related AEs
Description: Dose limiting toxicity (DLT) as defined by non-hematologic clinically significant grade 3 or 4 treatment-related AEs or hematologic grade 3 or 4 treatment related AEs that are clinically significant during the first cycle, graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE), Version 5.0.
Time Frame: Up to 24 months after treatment
Population: Per the protocol, this outcome measure specifically pertains to Phase I and, therefore, does not include Phase II participants. All Phase I participants were analyzed for this outcome. This clinical trial was terminated prematurely due to MEI Pharma's withdrawal of funding, which included discontinuation of participant follow-up. This analysis is based on limited data collected prior to discontinuation before reaching the intended endpoint.
Measure: Number; unit: Adverse events
Arm/Group | Phase I: ME-401 + R-CHOP Dose Level 1 | Phase I: ME-401 + R-CHOP Dose Level 2 | Phase II: ME-401 + R-CHOP
Number analyzed (Participants) | 3 | 6 | 0
Adverse events | 2 | 3 |

2. Primary Outcome: Phase II: Progression Free Survival (PFS) Assessed by Lugano Criteria
Description: PFS, as defined as time from study treatment initiation to documented disease progression per Lugano Criteria, or death from any cause, whichever occurs first.
Time Frame: 24 months (2 years)
Population: This clinical trial was terminated prematurely due to MEI Pharma's withdrawal of funding, which included discontinuation of participant follow-up. This analysis is based on limited data collected prior to discontinuation before reaching the intended endpoint. One participant in Phase II did not meet the protocol criteria for outcome analysis and is therefore excluded from this analysis.
Measure: Mean (Full Range); unit: months
Groups:
- Phase II: ME-401 + R-CHOP Dose Level 2; Phase II: ME-401 + R-CHOP: Participants will receive ME-401 dose dependent on dose-escalation schedule at time of enrollment - all will receive standard dose R-CHOP. ME-401 (60 mg) will be given on days 1-7 (dose level 2) of a 21 day cycle with standard dose R-CHOP x 6 cycles.
Arm/Group | Phase I: ME-401 + R-CHOP Dose Level 1 | Phase II: ME-401 + R-CHOP Dose Level 2 | Phase II: ME-401 + R-CHOP
Number analyzed (Participants) | 0 | 0 | 3
months |  |  | 5 [5 to 5]

3. Secondary Outcome: Phase I: Number of Treatment-related AEs
Description: Number of treatment-related AEs in Phase I.
  Participants will be followed for toxicity for 30 days after treatment has been discontinued or until death, whichever occurs first. The clinical course of each event will be followed until resolution, stabilization, or until it has been determined that the study treatment or participation is not the cause with a cut off of 24 months after completion of therapy.
Time Frame: Up to 24 months after treatment
Population: Per the protocol, this outcome measure pertains to Phase I and does not include Phase II participants. All Phase I participants were analyzed for this outcome. This clinical trial was terminated prematurely due to MEI Pharma's withdrawal of funding, which included discontinuation of participant follow-up. This analysis is based on limited data collected prior to discontinuation before reaching the intended endpoint.
Measure: Number; unit: adverse events
Arm/Group | Phase I: ME-401 + R-CHOP Dose Level 1 | Phase I: ME-401 + R-CHOP Dose Level 2 | Phase II: ME-401 + R-CHOP
Number analyzed (Participants) | 3 | 6 | 0
adverse events | 7 | 18 |

4. Secondary Outcome: Phase II: Number of Treatment-related AEs
Description: Number of treatment-related AEs in Phase II
  Participants will be followed for toxicity for 30 days after treatment has been discontinued or until death, whichever occurs first. The clinical course of each event will be followed until resolution, stabilization, or until it has been determined that the study treatment or participation is not the cause with a cut off of 24 months after completion of therapy.
Time Frame: Up to 24 months after treatment
Population: Per the protocol, this outcome measure pertains to Phase II and does not include Phase I participants. All Phase II participants were analyzed for this outcome. This clinical trial was terminated prematurely due to MEI Pharma's withdrawal of funding, which included discontinuation of participant follow-up. This analysis is based on limited data collected prior to discontinuation before reaching the intended endpoint.
Measure: Number; unit: treatment related adverse events
Arm/Group | Phase I: ME-401 + R-CHOP Dose Level 1 | Phase I: ME-401 + R-CHOP Dose Level 2 | Phase II: ME-401 + R-CHOP
Number analyzed (Participants) | 0 | 0 | 3
treatment related adverse events |  |  | 22

5. Secondary Outcome: Phase II: Number of Days Treatment is Delayed
Description: Number of days treatment is delayed
Time Frame: Up to 24 months after treatment
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Phase I: ME-401 + R-CHOP Dose Level 1 | Phase I: ME-401 + R-CHOP Dose Level 2 | Phase II: ME-401 + R-CHOP
Number analyzed (Participants) | 0 | 0 | 3
days |  |  | 0 (0)

6. Secondary Outcome: Phase II: Overall Response (OR) Assessed by Lugano Criteria
Description: OR assessed by Lugano criteria. OR is defined as achieving either CR or PR at any stage from time of commencement of protocol treatment to time of treatment cessation for whatever reason
Time Frame: 24 months (2 years)
Population: Per the protocol, this outcome measure pertains to Phase II and does not include Phase I participants. One participant in Phase II did not meet the protocol criteria for outcome analysis and is therefore excluded from this analysis. This clinical trial was terminated prematurely due to MEI Pharma's withdrawal of funding, which included discontinuation of participant follow-up. This analysis is based on limited data collected prior to discontinuation before reaching the intended endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I: ME-401 + R-CHOP Dose Level 1 | Phase I: ME-401 + R-CHOP Dose Level 2 | Phase II: ME-401 + R-CHOP
Number analyzed (Participants) | 0 | 0 | 3
Participants |  |  | 3

7. Secondary Outcome: Complete Response (CR) Assessed by Lugano Criteria
Description: CR assessed by Lugano criteria
Time Frame: 24 months (2 years)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I: ME-401 + R-CHOP Dose Level 1 | Phase I: ME-401 + R-CHOP Dose Level 2 | Phase II: ME-401 + R-CHOP
Number analyzed (Participants) | 0 | 0 | 3
Participants |  |  | 2

8. Secondary Outcome: Partial Response (PR) Assessed by Lugano Criteria
Description: PR assessed by Lugano criteria
Time Frame: 24 months (2 years)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I: ME-401 + R-CHOP Dose Level 1 | Phase I: ME-401 + R-CHOP Dose Level 2 | Phase II: ME-401 + R-CHOP
Number analyzed (Participants) | 0 | 0 | 3
Participants |  |  | 1

9. Secondary Outcome: Phase II: Duration of Response (DoR)
Description: DoR defined as the time from documented response (CR or PR) to the time of confirmed disease progression or death due to any cause, whichever occurs first
Time Frame: 24 months (2 years)
Population: Per the protocol, this outcome measure pertains to Phase II and does not include Phase I participants. One participant in Phase II did not meet the protocol criteria for outcome analysis and is therefore excluded from this analysis. This clinical trial was terminated prematurely due to MEI Pharma's withdrawal of funding, which included discontinuation of follow-up. This analysis is based on limited data (the average time from the participant's best response until discontinuation of follow-up).
Measure: Mean (Full Range); unit: months
Arm/Group | Phase I: ME-401 + R-CHOP Dose Level 1 | Phase II: ME-401 + R-CHOP Dose Level 2 | Phase II: ME-401 + R-CHOP
Number analyzed (Participants) | 0 | 0 | 3
months |  |  | 1 [0 to 2]

10. Secondary Outcome: Phase II: Overall Survival (OS)
Description: OS defined as the time from first dose of study treatment to death from any cause
Time Frame: 24 months (2 years)
Population: as for outcome 6
Measure: Mean (Full Range); unit: months
Arm/Group | Phase I: ME-401 + R-CHOP Dose Level 1 | Phase I: ME-401 + R-CHOP Dose Level 2 | Phase II: ME-401 + R-CHOP
Number analyzed (Participants) | 0 | 0 | 3
months |  |  | 5 [5 to 5]

11. Secondary Outcome: Phase II: Time to Treatment Failure
Description: Time to Treatment Failure defined as the time from study entry to any treatment failure.
Time Frame: 24 months (2 years)
Population: as for outcome 6
Measure: Mean (Full Range); unit: months
Arm/Group | Phase I: ME-401 + R-CHOP Dose Level 1 | Phase I: ME-401 + R-CHOP Dose Level 2 | Phase II: ME-401 + R-CHOP
Number analyzed (Participants) | 0 | 0 | 3
months |  |  | 5 [5 to 5]

ADVERSE EVENTS:
Time Frame: 24 months (2 years)
Arm/Group | Phase I: ME-401 + R-CHOP Dose Level 1 | Phase I: ME-401 + R-CHOP Dose Level 2 | Phase II: ME-401 + R-CHOP
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/6 | 0/4
Serious Adverse Events (participants affected / at risk) | 1/3 | 6/6 | 2/4
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I: ME-401 + R-CHOP Dose Level 1 (N=3) | Phase I: ME-401 + R-CHOP Dose Level 2 (N=6) | Phase II: ME-401 + R-CHOP (N=4)
Jejunal Perforation (Gastrointestinal disorders) | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 1 | 0
White blood cell count decreased (Investigations) | 1 | 2 | 0
Lung Infection (Infections and infestations) | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 0 | 1 | 0
Colonic obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 1
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I: ME-401 + R-CHOP Dose Level 1 (N=3) | Phase I: ME-401 + R-CHOP Dose Level 2 (N=6) | Phase II: ME-401 + R-CHOP (N=4)
Anemia (Blood and lymphatic system disorders) | 1 | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 2
Diarrhea (Gastrointestinal disorders) | 1 | 2 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 0
Fatigue (General disorders) | 0 | 2 | 1
Neutrophil count decreased (Investigations) | 1 | 0 | 0
White blood cell count decreased (Investigations) | 1 | 0 | 0
Platelet count decreased (Investigations) | 0 | 2 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0
Dysphasia (Nervous system disorders) | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Thromboembolic event (Vascular disorders) | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1
Alkaline phosphatase increased (Investigations) | 0 | 0 | 1
Lipase increased (Investigations) | 0 | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 1
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Upper respiratory infection (Infections and infestations) | 0 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
The pharmaceutical company, MEI Pharma, withdrew funding, therefore leading to a premature termination and follow-up was discontinued for all patients. All outcome analyses are based on only a small number of participants that were followed for a short period of time.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-04-22): https://cdn.clinicaltrials.gov/large-docs/35/NCT04517435/Prot_SAP_000.pdf
  • Informed Consent Form (2022-08-04): https://cdn.clinicaltrials.gov/large-docs/35/NCT04517435/ICF_001.pdf